CLINICAL TRIAL: NCT05402618
Title: Minimally Invasive Versus Open Surgery for Perihilar Cholangiocarcinoma(PHC)：A Multicenter Real-world Study
Brief Title: Minimally Invasive Versus Open Surgery for PHC
Status: Completed | Type: Observational
Sponsor: Renyi Qin (Other)
Responsible Party: Sponsor-Investigator, Renyi Qin, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJDBPS10
Record Dates: First submitted 2022-05-26; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Perihilar Cholangiocarcinoma
Keywords: laparoscopic; minimally invasive; open resection
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- minimally invasive surgery
  Interventions: Other: No intervention
- open surgery
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study without any intervention.

SUMMARY:
Brief Summary: This is a multicentric, retrospective, real-world study to investigate the surgical outcomes of minimally invasive surgery compared with open surgery for Perihilar Cholangiocarcinoma (PHC), with the perioperative characteristics and long-term overall survival being compared. We aimed to find out whether the minimally invasive surgery is safe or feasible for PHC. And we also want to find out patients with what kind of characteristic can be benefit from the minimally invasive surgery compared with the open approach.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed PHC.

Exclusion Criteria:

1. Peritoneal seeding or metastasis to the liver, para-aortic lymph nodes, or distant sites;
2. Non-adenocarcinoma histology;
3. Incomplete clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective review of a real-world institutional databases from 10 hospitals in China identified PHC patients who underwent curative LS or OP surgery (including R0 and R1) form January 2012 and January 2019.Patients with pathologically confirmed PHC and without any evidence of distant metastasis by preoperative examinations were included.
Sampling Method: Non-Probability Sample
Enrollment: 783 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative length of stay | up to 90 days
  defined as the time from being admitted to hospital to discharge
Overall survival | through study completion, an average of 5 year
  defined as the duration from the first day after surgery to either the date of death or the last follow-up

SECONDARY OUTCOMES:
Operation time | intraoperative
  defined as the time from skin incision or trocar placement to complete skin closure
postoperative complications | up to 90 days
  Postoperative complications were reviewed within 90 days after surgery and graded according to Clavien-Dindo (CD) classification system.Postoperative biliary leakage, hemorrhage, and liver failure were defined and classified according to the criteria set out by the International Study Group of Liver Surgery (ISGLS). Wound infection was defined as purulent drainage from the incision or/and positive findings of culture of the fluid or tissue aseptically obtained from the incision.
Reoperation within 90 days | up to 90 days
  defined as any reoperation within 90 days
Mortality | up to 90 days
  defined as any death within 30 days and 90 days, respectively
Readmission within 90 days | up to 90 days
  defined as any readmission within 90 days
Operative details | intraoperative
  including blood transfusion, vascular resection, number of resected lymph nodes
R0 resection | intraoperative
  defined as tumor-free margins in all the reported surgical margins (biliary and circumferential margins)
Intraoperative blood loss | intraoperative
  recorded by the anesthetist using a vacuum system
Vessel reconstruction | intraoperative
  defined as any repair or replacement of major vessels during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biliary and Pancreatic Surgery, Tongji Hospital, Affiliated Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Wang M, Qin T, Zhang H, Li J, Deng X, Zhang Y, Zhao W, Fan Y, Li D, Chen X, Feng Y, Zhu S, Xing Z, Yu G, Xu J, Xie J, Dou C, Ma H, Liu G, Shao Y, Chen W, Liu J, Liu J, Yin X, Qin R. Laparoscopic versus open surgery for perihilar cholangiocarcinoma: a multicenter propensity score analysis of short- term outcomes. BMC Cancer. 2023 May 3;23(1):394. doi: 10.1186/s12885-023-10783-9. PMID 37138243